CLINICAL TRIAL: NCT01207856
Title: Randomised Controlled Clinical Trial of Cognitive Rehabilitation in Multiple Sclerosis and Assessment by Neuroimaging
Brief Title: Randomised Controlled Clinical Trial of Cognitive Rehabilitation in Multiple Sclerosis
Acronym: REACTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Merck Serono International SA (Industry); ARSEP foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2010/07
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis; Cognitive Rehabilitation
Keywords: Multiple sclerosis; functional MRI; cognitive rehabilitation; ecological evaluation; neuroplasticity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group A (Active Comparator): specific cognitive rehabilitation
  Interventions: Behavioral: specific cognitive rehabilitation
- Groupe B : non specific rehabilitation (Active Comparator)
  Interventions: Behavioral: non specific cognitive rehabilitation
- group C (Other): group C for MRI, neuropsychological and ecological assessments
  Interventions: Other: no intervention

INTERVENTIONS:
Behavioral: specific cognitive rehabilitation — Individual rehabilitation procedures will be focused on attention, executive functions, IPS and working memory. The program will be tailored to each patient cognitive status depending on the impairments identified during the initial assessment while maintaining a systematic work on attention and executive functions. A total of 50 sessions lasting one hour at a rate of 3 sessions per week for a total period of 4 months will be proposed. Sessions will include varied exercises according to complexity and presentation modality, using computerized and "paper-and-pencil" tasks and metacognitive training. Work will be progressive, depending on the progresses achieved (increase complexity and intensity of the exercises according to success at the previous level of exercises).
  Arms: group A
Behavioral: non specific cognitive rehabilitation — A total of 50 sessions lasting one hour at a rate of 3 sessions per week for a total period of 4 months will be proposed by group composed to 5 patients
  Arms: Groupe B : non specific rehabilitation
Other: no intervention — no intervention
  Arms: group C

SUMMARY:
Despite the need for cognitive rehabilitation, there is a paucity of well-designed research studies to investigate treatment approaches or their effectiveness in MS. Most of published studies suffer from significant methodological flaws including small sample size, short follow-up periods, and lack of specific outcome criteria to determine improvement. O'Brien et al. (2008) recently reviewed 16 studies of cognitive rehabilitation designed to persons with MS and found only 4 class I studies and only one class I study of rehabilitation of attention deficits. Methodologically rigorous research is needed to confirm the preliminary results reported by these studies and determine the effectiveness and efficacy of cognitive rehabilitation interventions in attention deficits in MS. O'Brien et al. listed limitations found in previous studies that must be addressed in future studies. The present study was designed according to these recommendations. It is a randomized, controlled study, in parallel groups, evaluator blinded.

Number of participants: 25 RRMS patients in the active group, 25 RRMS patients in the control group and 25 healthy subjects.

The protocol will be proposed to RRMS patients AFFILIATED TO FRENCH SOCIAL SECURITY referred to the investigators center by practicing neurologists and fulfilling the inclusion criteria for screening.

Patients will be randomised between two groups. The active group (25 patients) will be treated by rehabilitation. Individual rehabilitation procedures will be focused on attention, executive functions and IPS. The program will be tailored to each patient cognitive status depending on the impairments identified during the initial assessment while maintaining a systematic work on attention and executive functions. A total of 50 sessions lasting one hour at a rate of 3 sessions per week for a total period of 4 months will be proposed. Patients randomized in the other group will participate to group session every week without specific cognitive rehabilitation. 25 healthy control subjects (group C), matched to patients for education, gender and age with patients of groups A/B will have the same evaluation procedures than patients.

Evaluation will be performed at baseline, after 4 months (end of treatment period) and after 8 months. Evaluation will include clinical testing, cognitive battery (paper/pencil and computer tests), cognitive ecological evaluation (Computer test of attention in a virtual reality environment and driving test on a driving simulator), questionnaires about daily life and MRI (fMRI and MRI). All patients and healthy subjects will undergo the fMRI protocol using a paradigm previously published by the investigators group (Bonnet et al., 2009): Go/No-go paradigm with increasing difficulty during four successive conditions (the Tonic Alertness task, Go/No-go (IG), reversal Go/No-go (RG), and complex Go/No-go (CG). In a previous study the investigators observed compensatory activation in MS patients as compared to healthy controls for the three first conditions and a saturation of compensatory processes for the more complex. In the present study, the investigators hypothesize that a similar pattern will occur at baseline and that cognitive rehabilitation will improve brain compensation at the fourth level of complexity.

DETAILED DESCRIPTION:
: Multiple Sclerosis (MS) is the most frequent disabling neurological disease in young adults. Over the past two decades, cognitive impairment in MS has received increasing interest. Although for a long time described in MS text books, it has been underestimated until recently. It is now accepted as an important feature of MS with a high impact on working and social abilities. The cognitive disorders in MS are dominated by a slowdown in information processing speed (IPS), as well as disturbances of attention and memory. The nature of cognitive findings suggest that the impairments depend on the integrity of large-scale cortical integrative processes, which involve long-distance white matter projections which can be impaired due to diffuse demyelinating injury in patients with MS. At the early stages of MS there is increasing evidence that neuroplasticity, the ability of the brain to respond to various insults, allows adaptive reorganization of cognitive functions to limit impairment, despite widespread tissue damage. Recently, we showed that at the early stages of RRMS compensatory capacities are relatively maintained, especially in highly-educated patients suggesting that cognitive training might be useful. The requirement of cerebral compensatory mechanisms to perform the cognitive tests was postulated in MS patients on the basis of functional MRI (fMRI) studies. By using a go/no go task of increasing complexity in a fMRI study in RRMS patients, we observed that a limitation of this compensatory cerebral recruitment appears when the attentional solicitations reach a particular level of difficulty. We postulate that a cognitive training program may help to maintain these compensatory capacities. Therefore, we propose to evaluate the effect of the program on brain activation using a task with several levels of attention requirement (increased attention load) by using fMRI and to evaluate in parallel its clinical effect and its impact in daily activities.

ELIGIBILITY:
Inclusion Criteria:

patients

* male or female relapsing remitting or secondary progressive or primary progressive Multiple sclerosis patients according to Polman et al. (2005),
* age 18-55; disease duration >6 months and ≤15 years,
* right handed,

Patients will be eligible for randomization (cognitive inclusion criterion) if they performed worse than :

* 2 scores <1 standard deviation (SD) on the scores evaluating information processing speed and attention (IPS-Attention) and 1 score <1DS on other tests assessing executive functions (EF) and working memory (WM).

or

* if they performed worse than 2 scores <1 SD on the 5 tests of information processing speed, attention and executive function (SDMT, Stroop and TMT battery GREFEX, and divided attention substests (TAP) and 1 score <1DS on other tests assessing information processing speed, and executive and attention functions (IPS / FAE) and working memory (WM).

healthy volunteers

* male or female,
* age 18-55 matched for age, gender and education
* Accepting to participate and signing the informed consent
* affiliated to french social security

Exclusion Criteria:

* existing other neurological or psychiatric disorder, visual, oculomotor, auditory and motor impairments precluding ability to perform computerized tasks and the driving simulator tasks,
* prior history of addictive behaviour,
* MS attack in the 2 months preceding the screening,
* corticosteroid pulse therapy within 2 months preceding screening,
* severe cognitive deficits or dementia (MMS<27), moderate to severe visuospatial incapacity (type IV or V at the Rey figure score < 28), moderate to severe depression (BDI >27),
* Participant without driving licence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Comparison between groups concerning the z cognitive global executive z score . | after 4 months (M4)

SECONDARY OUTCOMES:
Comparison of brain activation in the treated group versus control group at the fourth condition. | 4 and 8 months
Comparison between groups concerning the z score of the SDMT | 4 and 8 months
Comparison between groups of the daily-life cognitive questionnaire scores | at M4 and M8
Comparison between groups concerning the z cognitive global executive z score | 8 months
Clinical Global impression of patients | 4 and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Brochet, Md PhD, Study Director — University Hospital, Bordeaux
Locations (1):
- Service de Neurologie - Pôle des Neurosciences Cliniques, CHU de Bordeaux., Bordeaux, France

REFERENCES:
- [Derived] Moroso A, Ruet A, Lamargue-Hamel D, Munsch F, Deloire M, Coupe P, Ouallet JC, Planche V, Moscufo N, Meier DS, Tourdias T, Guttmann CR, Dousset V, Brochet B. Posterior lobules of the cerebellum and information processing speed at various stages of multiple sclerosis. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):146-151. doi: 10.1136/jnnp-2016-313867. Epub 2016 Oct 27. PMID 27789541